CLINICAL TRIAL: NCT00487630
Title: A Multicenter, Phase 4, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Recombinant Alpha-Galactosidase A (Agalsidase Beta, FABRAZYME) in Heterozygous Females for Fabry Disease
Brief Title: Evaluation of Efficacy and Safety of Agalsidase Beta in Heterozygous Females for Fabry Disease
Acronym: HEART
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM-01-076; PHRC National 2001
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-06

CONDITIONS: Fabry Disease
Keywords: Heterozygous females; Cardiomyopathy
MeSH Terms: conditions — Fabry Disease; Cardiomyopathies | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: recombinant alpha-galactosidase A

SUMMARY:
Fabry disease (OMIM 301500) is an X-linked inborn error of sphingolipid metabolism resulting from the deficiency of the lysosomal enzyme alpha-galactosidase A. Heterozygous females for Fabry disease may be symptomatic with cardiac, renal or cerebrovascular involvement. Clearance of Gb3 and stabilization of renal function has been demonstrated in male patients treated with agalsidase beta (FABRAZYME). In contrast, no randomized, controlled study of the efficacy of recombinant alpha-galactosidase A has been reported in heterozygotes for Fabry disease.

DETAILED DESCRIPTION:
The primary objective is to evaluate cardiac left ventricular mass (measured with echocardiography by unique investigator) in females over 15 years of age affected with Fabry disease receiving 70 mg of agalsidase beta every other week, as compared with an untreated controlled group matched for gender and age.

The secondary objectives include evaluation of :

* left ventricular posterior wall thickness (echocardiography)
* interventricular septum thickness (echocardiography)
* tissue doppler imaging (myocardial function)
* EKG
* creatinaemia
* serum cystatin C level
* urinary protein/creatinine ratio
* microalbuminuria
* Gb3 urinary levels

Evaluation of tolerance and safety with :

* Home therapy infusions follow up
* Vitals
* Physical examination
* Adverse events
* Antibodies levels

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 15 years with clinical and biological evidence of Fabry disease (GLA gene mutation detected)

Exclusion Criteria:

* Pregnancy
* Allergy to agalsidase beta
* Congestive heart failure
* Creatinaemia > 135 µmol/l
* Medical history of stroke during the last year
* Medical history of more than 2 transient ischemic attack
* Blood pressure > 160/95
* Modification in medications treating for blood pressure during the last 3 months before enrollment
* Complete absence of clinical or biological symptoms
* Weight > 87 kg or < 35 kg

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2005-06; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass | 2 years

SECONDARY OUTCOMES:
Posterior wall thickness, interventricular thickness, ECG, creatinaemia, urinary protein / creatinine ratio, microalbuminuria, urinary Gb3 level | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique P GERMAIN, MD, PhD, Principal Investigator — Centre de reference de la maladie de Fabry et des maladies hereditaires du tissu conjonctif. Assistance Publique Hopitaux de Paris
Locations (1):
- Centre de reference de la maladie de Fabry et des maladies hereditaires du tissu conjonctif. Assistance Publique - Hôpitaux de Paris, Paris, France